CLINICAL TRIAL: NCT02385474
Title: Effectiveness of Silver Diamine Fluoride in Arresting Dental Caries in Preschool Children: a Randomized Clinical Trial With Different Periodicity and Concentration.
Brief Title: Effectiveness of SDF in Arresting Dental Caries in Preschool Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU765213M
Record Dates: First submitted 2015-02-04; First posted 2015-03-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Early Childhood Caries
Keywords: silver diamine fluoride; randomized clinical trial; caries; children; fluoride
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 38% SDF semi-annual (Experimental): semi-annual application of 38% SDF
  Interventions: Drug: 38% SDF
- 38% SDF annual (Experimental): annual application of 38% SDF
  Interventions: Drug: 38% SDF
- 12% SDF semi-annual (Active Comparator): semi-annual application of 12% SDF
  Interventions: Drug: 12% SDF
- 12% SDF annual (Active Comparator): annual application of 12% SDF
  Interventions: Drug: 12% SDF

INTERVENTIONS:
Drug: 12% SDF — 12% silver diamine fluoride solution, of which the capability of arresting dental caries is not sure
  Other Names: 12% silver diamine fluoride
  Arms: 12% SDF annual; 12% SDF semi-annual
Drug: 38% SDF — 38% silver diamine fluoride solution, of which the capability of arresting dental caries is known
  Other Names: 38% silver diamine fluoride
  Arms: 38% SDF annual; 38% SDF semi-annual

SUMMARY:
Background: Tooth decay in children (Early childhood caries, or ECC) is a common childhood disease. Poor dentition significantly affects the nutrition, growth, development and general health of children. Conventional dental care for ECC is neither affordable nor accessible, particularly for the disadvantaged communities. Silver diamine fluoride (SDF) is a safe, cost-effective caries-arresting agent that appears to conform to the World Health Organization's Millennium Goals. SDF is commercially available at 38% and 12%, and topically used yearly or half-yearly to arrest ECC. The SDF regimens used for ECC treatment lack an evidence base. Therefore it is necessary to find the most suitable SDF concentration and application interval to arrest ECC. The purpose of this randomised controlled trial is to compare the efficacy of two commercially available SDF solutions at pre-prepared concentrations of 38% and 12% when applied at yearly or half-yearly intervals over 36 months in arresting caries in primary teeth.

Methods / Design: This double-blinded study has recruited 888 kindergarten children aged 3-4 years with caries. The sample size is sufficient for the appropriate statistical analyses. The children were classified into high and low caries rates and equally allocated into four groups for the caries treatment:

Group A - semi-annual application of 12% SDF; Group B - annual application of 12% SDF; Group C - semi-annual application of 38% SDF; Group D - annual application of 38% SDF. The children will be followed for 36 months in their kindergartens until they enter primary school. Clinical examinations at 6-month intervals will be conducted to assess whether the caries are arrested. Information on confounding factors, such as oral hygiene habits and the use of other fluoride agents, will be collected through a parental questionnaire at the baseline and follow-ups.

Discussion: This study will help determine the most suitable SDF concentration and application interval to arrest caries in children. Because SDF use for caries arrest is painless, simple, and low-cost, it can be widely recommended and promoted for caries control in young children or those with difficulty accessing and affording conventional dental care. The applicability of the findings and their impact on public health would be immense.

ELIGIBILITY:
Inclusion Criteria:

The children included in the study should

1. aged 3-4 years who have tooth decay and are attending the first year of kindergarten,
2. be generally healthy,
3. have parental consent, and
4. have at least 1 tooth with untreated caries that extends into the dentine.

Exclusion Criteria:

* Children who are uncooperative and difficult to manage, have major systemic diseases, or are on long-term medication will be excluded.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 888 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change of the baseline number of soft (active) caries surfaces that become arrested (hardened) at 30-month follow-up | 30-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hung Chu, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Braga MM, Mendes FM, De Benedetto MS, Imparato JC. Effect of silver diammine fluoride on incipient caries lesions in erupting permanent first molars: a pilot study. J Dent Child (Chic). 2009 Jan-Apr;76(1):28-33. PMID 19341576
- [Background] Chu CH, Fung DS, Lo EC. Dental caries status of preschool children in Hong Kong. Br Dent J. 1999 Dec 11;187(11):616-20; discussion 605. doi: 10.1038/sj.bdj.4800347. PMID 16163284
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Lo EC, Chu CH, Lin HC. A community-based caries control program for pre-school children using topical fluorides: 18-month results. J Dent Res. 2001 Dec;80(12):2071-4. doi: 10.1177/00220345010800120901. PMID 11808764
- [Derived] Duangthip D, Fung MHT, Wong MCM, Chu CH, Lo ECM. Adverse Effects of Silver Diamine Fluoride Treatment among Preschool Children. J Dent Res. 2018 Apr;97(4):395-401. doi: 10.1177/0022034517746678. Epub 2017 Dec 13. PMID 29237131
- [Derived] Fung MHT, Duangthip D, Wong MCM, Lo ECM, Chu CH. Randomized Clinical Trial of 12% and 38% Silver Diamine Fluoride Treatment. J Dent Res. 2018 Feb;97(2):171-178. doi: 10.1177/0022034517728496. Epub 2017 Aug 28. PMID 28846469